CLINICAL TRIAL: NCT07077200
Title: Comparison of Intranasal Dexmedetomidine and Short Video Viewing in the Management of Preoperative Anxiety and Sedation in Pediatric Endoscopy
Brief Title: Comparison of Intranasal Dexmedetomidine and Short Video Viewing in the Preoperative Anxiety
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, caner genc, Associate professor (Anesthesiology Specialist), Samsun University
Other Study IDs: Intranasal Dex Vs Short Videos
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia; Sedation; Anxiety
Keywords: Intranasal dexmedetomidine; Non-operating room anesthesia; Preoperative anxiety; Pediatric endoscopy; Short video viewing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- İntranasal Dexmedetomidine: Patients will be admitted to the preoperative holding area prior to the procedure. Upon arrival, intranasal dexmedetomidine will be administered at a dose of 3 mcg/kg via a mucosal atomiser device. The Modified Yale Preoperative Anxiety Scale (mYPAS) will be used to assess anxiety levels at three time intervals: upon arrival in the procedure room, immediately before transfer to the procedure room, and at the initiation of sedoanalgesia (induction).
  Interventions: Other: Intranasal dexmedetomidine
- Short videos: Patients will be admitted to the preoperative holding area prior to the procedure. The Modified Yale Preoperative Anxiety Scale (mYPAS) will be used to assess anxiety levels at the following time points: upon arrival in the holding area, immediately before transfer to the procedure room, and at the initiation of sedoanalgesia.
  In the waiting area, children will be allowed to watch short videos on a platform of their choice (e.g., YouTube Shorts, TikTok, Instagram Shorts, cartoons, etc.) using the phone or tablet they typically use at home with their families. All content will be filtered for child-appropriate material. Children who refuse to watch or encounter technical issues during the video session will be excluded from the study.

INTERVENTIONS:
Other: Intranasal dexmedetomidine — This intervention is distinguished by the use of intranasal dexmedetomidine at a standardized dose of 3 mcg/kg, administered non-invasively upon the child's arrival in the preoperative holding area. Unlike other pharmacological methods that often require intravenous access or oral administration, this approach minimizes procedural stress and discomfort, which is particularly advantageous in pediatric populations.
  Dexmedetomidine is a selective alpha-2 adrenergic agonist known for its anxiolytic, sedative, and analgesic properties, without causing significant respiratory depression-a key concern with agents like benzodiazepines or opioids. Its intranasal delivery provides a rapid onset of action while maintaining hemodynamic stability, which is critical during the preoperative period.
  This intervention is also notable for its comparison with a non-pharmacological strategy-short video viewing-making the study unique in evaluating the relative efficacy of a low-risk pharmacologic option
  Groups: İntranasal Dexmedetomidine

SUMMARY:
This observational study aims to compare the effects of short video viewing and intranasal dexmedetomidine administration-both of which are part of routine clinical practices in the pediatric endoscopy unit-on preoperative anxiety levels and the need for intravenous sedation. Patients who are exposed to these interventions as part of routine clinical care will be included in the study.

DETAILED DESCRIPTION:
Pediatric patients scheduled for upper or lower gastrointestinal endoscopy in the hospital's endoscopy unit and who receive either short video viewing or intranasal dexmedetomidine as part of standard clinical practice will be included in this study. The primary objective is to compare these two modalities in terms of preoperative anxiety, requirement for sedative agents, difficulty of intravenous access, and levels of satisfaction reported by parents and endoscopists.

This study will be conducted with a prospective and observational design. Preoperative anxiety levels will be assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS) at three distinct time points:

T1: Upon arrival in the preoperative holding area, T2: Prior to transfer to the endoscopy suite, T3: immediately before anesthesia induction. The consumption of sedative agents (e.g., propofol) will be recorded in terms of total dosage (mg) and dosage per kilogram of body weight (mg/kg). The difficulty of intravenous access will be rated on a 5-point scale. Parental satisfaction will be assessed using the PedsQL Healthcare Satisfaction Scale, while endoscopist satisfaction will be evaluated using a 5-point Likert scale. Statistical analyses will be performed to compare the outcomes between the two study groups.

Short Video Viewing Group:

All patients will be brought to the preoperative preparation area. Anxiety assessments using the mYPAS will be conducted at the designated time points. Patients will be allowed to watch short videos (such as YouTube Shorts, TikTok, Instagram Shorts, or cartoons), selected based on their preferences and filtered for age-appropriateness. Patients who refuse to watch the videos or encounter technical difficulties will be excluded from the study.

Intranasal Dexmedetomidine Group:

Patients in this group will receive intranasal dexmedetomidine via a mucosal atomiser device at a dose of 3 mcg/kg upon arrival at the preoperative holding area. mYPAS assessments will be carried out at the same three time points.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 2-12 years undergoing endoscopy and/or colonoscopy, classified as ASA I-II

Exclusion Criteria:

* Patients under 2, over 12, or with ASA score >2
* Epilepsy
* Cardiovascular diseases
* Refuse to participate

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study included patients aged 2-12 years, classified as ASA I-II, who were scheduled to undergo endoscopy and/or colonoscopy by a pediatric gastroenterologist based on a clinical indication
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (mYPAS) scores | 1hour
  Preoperative anxiety levels will be assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS) at three distinct time points:
  T1: upon arrival in the preoperative holding area, T2: prior to transfer to the endoscopy suite, T3: immediately before anesthesia induction.

SECONDARY OUTCOMES:
Recovery Time | 1 hour
  The duration of patient monitoring in the recovery unit continued until a Modified Aldrete Score of 9 or higher was achieved.
Sedation Scores | 2 hour
  Sedation levels assessed using the Ramsay Sedation Scale (RSS) in the preoperative preparation unit, procedure room, and recovery unit constituted the secondary outcome of the study.
The difficulty level of intravenous (IV) access | 1 hour
  "The difficulty level of intravenous (IV) access was assessed using a 5-point Likert scale.
Endoscopist satisfaction | 2 hour
  Endoscopist satisfaction was evaluated with a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Caner Genc, M.D., Principal Investigator — Samsun University
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turunc E, Ustun YB, Bilgin S, Kaya C, Koksal E, Dost B. Effect of nebulized dexmedetomidine on gag reflex suppression and sedation quality in pediatric patients undergoing gastrointestinal endoscopy: a randomized controlled trial. BMC Anesthesiol. 2025 May 3;25(1):227. doi: 10.1186/s12871-025-03106-x. PMID 40319232